CLINICAL TRIAL: NCT06312995
Title: Pre-market Clinical Investigation of a Medical Device for the Immobilisation of Radius and Ulna Fractures in Paediatric Patients
Brief Title: Investigation of a Medical Device for the Immobilisation of Radius and Ulna Fractures in Paediatric Patients
Acronym: T3DDY02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Alessandro Zanardi, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: T3DDY02
Record Dates: First submitted 2024-02-13; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone | interventions — Casts, Surgical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T3DDY01 (Experimental): Acquired a digital acquisition of the patient's forearm using the Intel RealSense D415. The arm of the patient' is placed on a support to allow the plaster nurse to position of the wrist at the correct angle to treat the fracture. The limb is temporarily immobilised in a plaster cast by the nurses of the practice. The patient is booked for a subsequent outpatient visit (which will be conducted within 72 hours of digital acquisition of the forearm) for the application of the device under investigation. The production of the device through a Stratasys F370 3D printer owned by the Meyer Children's Hospital IRCCS. The material used is ABS (Acrylonitrile butadiene styrene) supplied by Stratasys and specific to the machine. Placement of the device on the patient by the investigating nurses, after removal of the temporary device. Collection of data on the evaluation of study parameters.
  Interventions: Device: T3DDY01
- PLASTER (Active Comparator): Traditional device placement (antibrachio-metacarpal cast). Radiological check at 7 days after trauma to verify the angle of the stumps fracture angle, followed by radiological check at 14 days if necessary . Removal of the plaster cast 30 days after the trauma, radiological check to verify the formation of bone callus, clinical evaluation and data collection at the end of treatment
  Interventions: Device: PLASTER

INTERVENTIONS:
Device: T3DDY01 — Digital acquisition of the patient's forearm using Intel RealSense D415 cameras (CE devices certified according to EN/IEC 60825-1 2007 - Safety of Laser product as Class I Laser Devices, i.e., Non-Hazardous Laser Radiation). The patient's arm is placed on a support to allow the plaster nurse to position the wrist at the correct angle needed to treat the fracture.
  Arms: T3DDY01
Device: PLASTER — Standard treatment plaster for fractures.
  Arms: PLASTER

SUMMARY:
Single-centre, randomised, controlled, non-profit study on a custom-made medical device for immobilisation of radius and ulna fracture in paediatric patients.

The aim of the study is to evaluate the benefits in terms of comfort, safety and efficacy resulting from the use of a customised 3D-printed wrist immobilisation device in children aged between 7 and 13 with a fracture of the distal metaphysis of radius or ulna of the 'green stick' type, compared to a control group treated with traditional immobilisation devices. The patients will be randomised between use of customised 3D- printed wrist immobilisisation device and plaster.

DETAILED DESCRIPTION:
The device under investigation has already been the subject of a pilot study (clinical investigation code: T3DDY01) with significant result. These results are also preparatory to the proposed new investigation, which aims to extend its applicability to more complex clinical conditions. Compared to the previous one, the new study will be able to take advantage of an improved acquisition process of the anatomy of the child's upper limb, obtained by updating the model of the chambers used.

The aim of the study is to evaluate the benefits in terms of comfort, safety and efficacy resulting from the use of a customised 3D-printed wrist immobilisation device in children aged between 7 and 13 with a fracture of the distal metaphysis of radius or ulna of the 'green stick' type, compared to a control group treated with traditional immobilisation devices. The patients will be randomised between use of customised 3D- printed wrist immobilisisation device and plaster.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 7 and 13 years with compound fracture of the distal metaphysis of radius and/or ulna at "green wood" and initial angulation <20°;
* Informed consent obtained.

Exclusion Criteria:

* Complete fracture of radius and ulna;
* Open fracture of radius and ulna;
* Polytrauma, polyfracture;
* Presence of neurovascular deficit at presentation;
* Presence of underlying bone disease;
* Presence of acute or chronic skin disorders;
* Psycho-behavioural disorders;
* Presence of ≥1 skin lesions according to NPUAP/EPUAP classification;
* Specific allergies related to the materials used in the tested device;
* Inability to perform follow-up examinations.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Fracture Healing | At 7 and 30 day from the use of the device
  Completion of the therapeutic course, i.e. fracture healing without intervention following immobilisation device placement with residual angulation < 20°. Radiographic assessment of the fracture angle at 7 and 30 days after application of the device application;
  * Radiographic assessment of fracture healing at 30 days, defined as presence of bone callus on 3 out of 4 fracture margins;
  * If at the 7-day assessment the fracture angle appears critical, defined as >15° or an increase >5° from the initial radiograph, the patient will undergo a further radiographic assessment after a further 7 days (i.e. 14 days from the start of treatment).
  * Functional recovery of the limb will be investigated with a clinical examination 30 days after removal of the device (60 from the start of treatment), where arc of motion and elective pain and painability to active mobilisation, as per normal clinical practice.

SECONDARY OUTCOMES:
Adverse event | through study completetion, an average of 1 year
  Recording at each assessment time of any adverse events such as: mobilisation of the device, appearance of peripheral deficits, intolerance expressed by the patient towards the device.
Comfort of use of devices | During the study (at 7 and 30 days from the use of the device)
  Administration of the Comfort Rating Scale. The comfort rating scales (CRS) measure wearable comfort across 6 dimensions. These dimensions are Emotion, Attachment, Harm, Perceived change, Movement and Anxiety. Each parameter has a 21 point scale which are scored from 0 (low) to 20 (high)
  Emotion description: I am worried about how I look when I wear this device. I feel tense or on edge because I am wearing the device.
  Attachment description: I can feel the device on my body. I can feel the device moving.
  Harm description: The device is causing me some harm. The device is painful to wear.
  Perceived change description: Wearing the device makes me feel physically different. I feel strange wearing the device.
  Movement description: The device affects the way I move. The device inhibits or restricts my movement.
  Anxiety description: I do not feel secure wearing the device
Presence of skin lesions or other manifestations of intolerance to the device | During the tudy (at 30 days)
  Presence of skin lesions or other manifestations of intolerance to the device:
  scale NPUAP/EPUAP (European Pressure Ulcer Advisory Panel) at 30 days scale NPUAP/EPUAP : min(Category I: Non-bleaching erythema), max (Category IV: Full thickness tissue loss)
Pain evaluation | During the study (7, 30-day and FU)
  Pain assessment with VAS ( Visual Analogue Scale) scale at 7- and 30-day follow-up (FU)
  VAS SCALE: 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Acceptance of the device | At 7 and 30 days from the use of the device
  dedicated Likaert scale administered at 7 and 30 days, only to parents for patients < 10 years, to parents and patients for age > 10 years
  Likaert scale: measure opinions, attitudes, or behaviors. It consists of a statement or a question, followed by a series of five or seven answer statements
Structural analysis of devices | 30 days After the start of the treatment
  Structural analysis of the newly manufactured device and at the end of treatment: macroscopic visual analysis to assess the global and local integrity of the device, performed by study nurse.
Usability for design purposes of the controlate | Through study completion, an average of 1 year
  Usability for planning purposes of the contralateral anatomical segment: superposition of the two models (mirroring+recording) and calculation of the deviation as point-to-point distance

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Zanardi, MD, Principal Investigator — Meyer Children's Hospital IRCCS Locations: Italy
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy